CLINICAL TRIAL: NCT03550989
Title: Assessment of Passive Environmental Aerosol Exposure Through IQOS (Tobacco Heating System [THS] With Marlboro Heatsticks) in a Restaurant Setting Where IQOS Use, But Not Cigarette Smoking, is Allowed.
Brief Title: Real-Life Passive Exposure Assessment of IQOS
Status: Completed | Type: Observational
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: P1-PES-01-JP
Record Dates: First submitted 2018-03-20; First posted 2018-06-11 (Actual); Results first posted 2019-07-29 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Environmental Exposure
Keywords: Environmental Aerosol Exposure; Environmental Tobacco Smoke; Indoor Air Quality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-Smokers: Each participant can participate in one Non-Exposure Event and one Exposure Event only.
  * Abstinent for at least 12 months from the use of any nicotine and/or tobacco-containing product based on self-reporting.
  * Must not be exposed to tobacco or nicotine-containing products use in any other substantial way (family, partner, workplace, etc.).
  Interventions: Other: Non-Exposure Event; Other: Exposure Event
- Cigarette Smokers: Each participant can participate in one Non-Exposure Event and one Exposure Event only.
  * Used at least 100 cigarettes
  * Smokes cigarettes daily > 1/day
  * Uses IQOS less than daily
  * Uses less than 30 HeatSticks/month
  * Cigarette is > 95% of tobacco/nicotine product (all product use)
  Interventions: Other: Non-Exposure Event; Other: Exposure Event
- IQOS Passive Users (not using IQOS): Each participant can participate in one Non-Exposure Event and one Exposure Event only.
  * Used at least 100 HeatSticks
  * Uses IQOS daily > 1/day
  * Smokes a cigarette less than daily
  * Smokes less than 30 cigarettes/month
  * IQOS is > 95% of tobacco/nicotine product (all product use) - excluding other products (e-cig/Ploom/etc.)
  Interventions: Other: Non-Exposure Event; Other: Exposure Event
- IQOS Active Users (using IQOS): Each participant can participate in one Exposure Event only.
  * Used at least 100 HeatSticks
  * Uses IQOS daily > 1/day
  * Smokes a cigarette less than daily
  * Smokes less than 30 cigarettes/month
  * IQOS is > 95% of tobacco/nicotine product (all product use) - excluding other products (e-cig/Ploom/etc.)
  Interventions: Other: Exposure Event

INTERVENTIONS:
Other: Non-Exposure Event — Non-Exposure event of 4h duration for the individual participants, where no use of any tobacco or nicotine-containing product is allowed, designed to establish background measurements in the absence of exposure to IQOS.
  Groups: Cigarette Smokers; IQOS Passive Users (not using IQOS); Non-Smokers
Other: Exposure Event — Exposure Event designed to measure urinary BoExp to selected HPHCs representative of ETS in all participant groups, with up to 5h of exposure to IQOS tobacco environmental aerosol for non-smokers, cigarette smokers (not using any tobacco or nicotine-containing product, including cigarettes), and IQOS passive users (not using IQOS). Additionally, this event includes up to 8h of exposure for IQOS active users (using IQOS).

SUMMARY:
This study is a non-interventional observational study designed to assess the impact of passive exposure to IQOS environmental tobacco aerosol in Non-Smokers in a real-life restaurant setting.

DETAILED DESCRIPTION:
The purpose of the study is to show that Non-Smokers, exposed to environmental tobacco aerosol from IQOS in a restaurant setting, do not have higher urinary levels of Biomarkers of Exposure (BoExp) to selected Harmful and Potentially Harmful Constituents (HPHCs), representative of Environmental Tobacco Smoke (ETS), compared to the urinary levels of BoExp measured in Non-Smokers before IQOS environmental tobacco aerosol exposure.

Furthermore, the impact of passive exposure to IQOS environmental tobacco aerosol on IQOS Users and Cigarette Smokers, not using any tobacco or nicotine-containing products, will be investigated. This will enable the assessment of individuals with varying levels of exposure to HPHCs and determine whether there is any measurable additional exposure related to the environmental tobacco aerosol from IQOS.

The study will also evaluate Indoor Air Quality (IAQ) through the assessment of concentrations of nicotine and selected HPHCs representative of tobacco-specific and IAQ markers in the air during exposure and non-exposure periods in a real-life restaurant setting.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to understand the information provided in the Subject Information Sheet (SIS) and Informed Consent Form (ICF) (confirmed by signing the ICF) and has signed the ICF.
* Adults legally authorized to buy tobacco products in Japan (20 years of age).
* Participant is Japanese as self-reported.
* Willing to participate in the study, comply with study procedures and has access to the Internet.
* Participant is an active IQOS User, Cigarette smoker or Non-Smoker as self-reported

Exclusion Criteria:

* Participant with a medical history of severe cardiovascular or respiratory diseases (e.g., stroke, acute cardiovascular event, pulmonary thrombosis) in the last 12 months as self-reported.
* Participant with currently active cancer or history of cancer within the last 5 years as self-reported.
* Female participant who is pregnant or breast-feeding as self-reported.
* Participant is a current or former employee of the tobacco industry or their first-degree relatives (parent and child).
* Participant is an employee of Philip Morris International (PMI), an employee of the Contract Research Organization (CRO) engaged for this study, an employee of the CRO's vendors, an employee of the restaurant/event location, or their first-degree relatives (parent or child).

Exclusion criteria specific to participants who are Non-Smokers:

* Participant lives in a household with users of tobacco or nicotine-containing products, or is exposed to the use of tobacco or nicotine-containing products at the workplace.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female or male Japanese IQOS Users, Cigarette smokers, or Non-Smokers.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Picavet, MD, Study Chair — Philip Morris Products S.A.; Takao Ohki, MD, PhD, Principal Investigator — Jikei University School of Medicine, Tokyo
Locations (1):
- Angepatio Restaurant, Shibuya-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Smokers: Each participant can participate in one Non-Exposure Event and one Exposure Event only.
  * Abstinent for at least 12 months from the use of any nicotine and/or tobacco-containing product based on self-reporting.
  * Must not be exposed to tobacco or nicotine-containing products use in any other substantial way (family, partner, workplace, etc.).
  Non-Exposure Event: Non-Exposure event of 4h duration for the individual participants, where no use of any tobacco or nicotine-containing product is allowed, designed to establish background measurements in the absence of exposure to IQOS.
  Exposure Event: Exposure Event to measure urinary BoExp to selected HPHCs representative of ETS in all participant groups, with up to 5h of exposure for non-smokers, cigarette smokers (not using any tobacco or nicotine-containing product, including cigarettes), and IQOS passive users (not using IQOS). Additionally, this event includes up to 8h of exposure for IQOS active users (using IQOS).
- Cigarette Smokers: Each participant can participate in one Non-Exposure Event and one Exposure Event only.
  * Used at least 100 cigarettes
  * Smokes cigarettes daily > 1/day
  * Uses IQOS less than daily
  * Uses less than 30 HeatSticks/month
  * Cigarette is > 95% of tobacco/nicotine product (all product use)
  Non-Exposure Event: Non-Exposure event of 4h duration for the individual participants, where no use of any tobacco or nicotine-containing product is allowed, designed to establish background measurements in the absence of exposure to IQOS.
  Exposure Event: Exposure Event to measure urinary BoExp to selected HPHCs representative of ETS in all participant groups, with up to 5h of exposure for non-smokers, cigarette smokers (not using any tobacco or nicotine-containing product, including cigarettes), and IQOS passive users (not using IQOS). Additionally, this event includes up to 8h of exposure for IQOS active users (using IQOS).
- IQOS Passive Users (Not Using IQOS): Each participant can participate in one Non-Exposure Event and one Exposure Event only.
  * Used at least 100 HeatSticks
  * Uses IQOS daily > 1/day
  * Smokes a cigarette less than daily
  * Smokes less than 30 cigarettes/month
  * IQOS is > 95% of tobacco/nicotine product (all product use) - excluding other products (e-cig/Ploom/etc.)
  Non-Exposure Event: Non-Exposure event of 4h duration for the individual participants, where no use of any tobacco or nicotine-containing product is allowed, designed to establish background measurements in the absence of exposure to IQOS.
  Exposure Event: Exposure Event to measure urinary BoExp to selected HPHCs representative of ETS in all participant groups, with up to 5h of exposure for non-smokers, cigarette smokers (not using any tobacco or nicotine-containing product, including cigarettes), and IQOS passive users (not using IQOS). Additionally, this event includes up to 8h of exposure for IQOS active users (using IQOS).
- IQOS Active Users (Using IQOS): Each participant can participate in one Exposure Event only.
  * Used at least 100 HeatSticks
  * Uses IQOS daily > 1/day
  * Smokes a cigarette less than daily
  * Smokes less than 30 cigarettes/month
  * IQOS is > 95% of tobacco/nicotine product (all product use) - excluding other products (e-cig/Ploom/etc.)
  Exposure Event: Exposure Event to measure urinary BoExp to selected HPHCs representative of ETS in all participant groups, with up to 5h of exposure for non-smokers, cigarette smokers (not using any tobacco or nicotine-containing product, including cigarettes), and IQOS passive users (not using IQOS). Additionally, this event includes up to 8h of exposure for IQOS active users (using IQOS).
Period: Overall Study
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS)
Started | 190 | 74 | 77 | 60
Completed | 188 | 73 | 76 | 60
Not Completed | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Smokers: * Abstinent for at least 12 months from the use of any nicotine and/or tobacco-containing product based on self-reporting.
  * Must not be exposed to tobacco or nicotine-containing products use in any other substantial way (family, partner, workplace, etc.).
- Cigarette Smokers: * Used at least 100 cigarettes
  * Smokes cigarettes daily > 1/day
  * Uses IQOS less than daily
  * Uses less than 30 HeatSticks/month
  * Cigarette is > 95% of tobacco/nicotine product (all product use)
- IQOS Passive Users (Not Using IQOS); IQOS Active Users (Using IQOS): * Used at least 100 HeatSticks
  * Uses IQOS daily > 1/day
  * Smokes a cigarette less than daily
  * Smokes less than 30 cigarettes/month
  * IQOS is > 95% of tobacco/nicotine product (all product use)
  * excluding other products (e-cig/Ploom/etc.)
- Total: Total of all reporting groups
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS) | Total
Number analyzed (Participants) | 190 | 74 | 77 | 60 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (12.52) | 49.9 (14.40) | 43.6 (11.08) | 38.8 (11.00) | 44.4 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 10 | 21 | 13 | 121
  Male | 113 | 64 | 56 | 47 | 280
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese Origin | 190 | 74 | 77 | 60 | 401
Region of Enrollment [Number; unit: participants]
  Japan | 190 | 74 | 77 | 60 | 401

OUTCOME MEASURES:

1. Primary Outcome: NEQ: (Non-Exposure Event)
Description: To measure nicotine equivalents (NEQ, a biomarker of exposure to Nicotine): molar sum of free nicotine, nicotine-glucuronide, free cotinine, cotinine-glucuronide, free trans-3'-hydroxycotinine, trans-3'-hydroxycotinine-glucuronide in spot urine (expressed as concentration adjusted to creatinine).
Time Frame: Measured in a baseline urine sample collected before the start of the event and in a final urine sample taken prior to leaving the event (4h exposure, minimum 2h exposure).
Population: Some participants were excluded from analysis for protocol deviations (including but not limited to, missing questionnaires, attended events but was not eligible to attend, assigned to an incorrect group, or missing samples).
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS)
Number analyzed (Participants) | 77 | 32 | 32
mg/g
  Baseline: number analyzed (Participants) | 70 | 27 | 27
  Baseline | 0.03845 [0.03120 to 0.04739] | 4.159 [2.253 to 7.678] | 5.695 [4.286 to 7.567]
  Final void: number analyzed (Participants) | 73 | 30 | 31
  Final void | 0.06876 [0.05527 to 0.08553] | 5.175 [2.902 to 9.228] | 6.821 [5.127 to 9.074]

2. Primary Outcome: NEQ: (Exposure Event)
Description: To measure nicotine equivalents (NEQ, a biomarker of exposure to Nicotine): molar sum of free nicotine, nicotine-glucuronide, free cotinine, cotinine-glucuronide, free trans-3'-hydroxycotinine, trans-3'-hydroxycotinine-glucuronide in spot urine (expressed as concentration adjusted to creatinine), during exposure events where some subjects used IQOS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS)
Number analyzed (Participants) | 113 | 42 | 45 | 60
mg/g
  Baseline: number analyzed (Participants) | 112 | 38 | 44 | 59
  Baseline | 0.04078 [0.03397 to 0.04896] | 3.051 [1.720 to 5.414] | 5.277 [4.018 to 6.930] | 4.683 [3.553 to 6.171]
  Final void: number analyzed (Participants) | 112 | 42 | 45 | 60
  Final void | 0.06205 [0.05000 to 0.07700] | 2.889 [1.573 to 5.308] | 5.974 [4.696 to 7.598] | 8.499 [6.667 to 10.83]

3. Primary Outcome: Total NNAL: (Non-Exposure Event)
Description: To measure Total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (Total NNAL, a BoExp to Tobacco Specific Nitrosamines) in spot urine (expressed as concentration adjusted to creatinine).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS)
Number analyzed (Participants) | 77 | 32 | 32
ng/g
  Baseline: number analyzed (Participants) | 74 | 27 | 28
  Baseline | NA [NA to NA] — Below the limit of quantification. | 69.65 [46.62 to 104.0] | 20.55 [13.91 to 30.36]
  Final Void: number analyzed (Participants) | 75 | 26 | 31
  Final Void | NA [NA to NA] — Below the limit of quantification. | 81.64 [59.48 to 112.1] | 27.41 [18.88 to 39.80]

4. Primary Outcome: Total NNAL: (Exposure Event)
Description: To measure Total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (Total NNAL, a BoExp to Tobacco Specific Nitrosamines) in spot urine (expressed as concentration adjusted to creatinine), during exposure events where some subjects used IQOS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS)
Number analyzed (Participants) | 113 | 42 | 45 | 60
ng/g
  Baseline: number analyzed (Participants) | 113 | 38 | 44 | 59
  Baseline | NA [NA to NA] — Below the limit of quantification. | 48.57 [34.57 to 68.25] | 19.68 [15.78 to 24.56] | 21.50 [16.29 to 28.38]
  Final Void: number analyzed (Participants) | 113 | 42 | 45 | 58
  Final Void | NA [NA to NA] — Below the limit of quantification. | 58.74 [45.76 to 75.39] | 20.31 [15.83 to 26.06] | 30.45 [23.91 to 38.77]

5. Primary Outcome: Total NNN: (Non-Exposure Event)
Description: To measure Total N-nitrosonornicotine (Total NNN, a BoExp to Tobacco Specific Nitrosamines) in spot urine (expressed as concentration adjusted to creatinine).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS)
Number analyzed (Participants) | 77 | 32 | 32
ng/g
  Baseline: number analyzed (Participants) | 74 | 27 | 27
  Baseline | NA [NA to NA] — Below the limit of quantification. | 3.945 [2.885 to 5.392] | 1.493 [0.9808 to 2.272]
  Final Void: number analyzed (Participants) | 75 | 25 | 29
  Final Void | NA [NA to NA] — Below the limit of quantification. | 4.008 [2.395 to 6.708] | 3.093 [1.826 to 5.240]

6. Primary Outcome: Total NNN: (Exposure Event)
Description: To measure Total N-nitrosonornicotine (Total NNN, a BoExp to Tobacco Specific Nitrosamines) in spot urine (expressed as concentration adjusted to creatinine) during exposure events where some subjects used IQOS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS)
Number analyzed (Participants) | 113 | 42 | 45 | 60
ng/g
  Baseline: number analyzed (Participants) | 112 | 38 | 44 | 58
  Baseline | NA [NA to NA] — Below the limit of quantification. | 2.694 [1.843 to 3.939] | 1.753 [1.396 to 2.201] | 0.9088 [0.6614 to 1.249]
  Final Void: number analyzed (Participants) | 113 | 42 | 45 | 56
  Final Void | NA [NA to NA] — Below the limit of quantification. | 3.992 [2.647 to 6.019] | 2.034 [1.333 to 3.104] | 2.347 [1.761 to 3.128]

7. Secondary Outcome: HPMA (Non-Exposure Events)
Description: To measure 3-hydroxy-1-methylpropylmercapturic acid (HMPMA, a BoExp to Crotonaldehyde ) in spot urine (concentration adjusted for creatinine).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS)
Number analyzed (Participants) | 77 | 32 | 32
μg/g
  Baseline: number analyzed (Participants) | 70 | 27 | 27
  Baseline | 103.2 [87.58 to 121.7] | 318.6 [249.4 to 406.9] | 133.2 [94.67 to 187.4]
  Final void: number analyzed (Participants) | 71 | 22 | 30
  Final void | 232.6 [191.1 to 283.0] | 307.7 [227.9 to 415.4] | 211.9 [160.4 to 280.0]

8. Secondary Outcome: HPMA (Exposure Events)
Description: To measure 3-hydroxy-1-methylpropylmercapturic acid (HMPMA, a BoExp to Crotonaldehyde ) in spot urine (concentration adjusted for creatinine), during exposure events where some subjects used IQOS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS)
Number analyzed (Participants) | 113 | 42 | 45 | 60
μg/g
  Baseline: number analyzed (Participants) | 112 | 38 | 43 | 59
  Baseline | 82.91 [74.36 to 92.44] | 233.4 [181.7 to 299.8] | 92.85 [82.83 to 104.1] | 103.0 [84.78 to 125.1]
  Final void: number analyzed (Participants) | 107 | 41 | 44 | 57
  Final void | 170.9 [152.4 to 191.7] | 224.1 [186.3 to 269.5] | 166.7 [137.3 to 202.4] | 195.3 [165.3 to 230.7]

9. Secondary Outcome: 3-HPMA (Non-Exposure Events)
Description: To measure 3 hydroxypropylmercapturic acid (3-HPMA, a BoExp to Acrolein) in spot urine (concentration adjusted for creatinine).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS)
Number analyzed (Participants) | 77 | 32 | 32
μg/g
  Baseline: number analyzed (Participants) | 70 | 27 | 27
  Baseline | 242.1 [207.6 to 282.5] | 935.7 [742.2 to 1180] | 454.9 [356.0 to 581.3]
  Final Void: number analyzed (Participants) | 70 | 22 | 29
  Final Void | 1108 [840.7 to 1461] | 1334 [950.9 to 1871] | 1240 [868.0 to 1771]

10. Secondary Outcome: 3-HPMA (Exposure Events)
Description: To measure 3 hydroxypropylmercapturic acid (3-HPMA, a BoExp to Acrolein) in spot urine (concentration adjusted for creatinine), during exposure events where some subjects used IQOS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS)
Number analyzed (Participants) | 113 | 42 | 45 | 60
μg/g
  Baseline: number analyzed (Participants) | 112 | 38 | 43 | 59
  Baseline | 246.6 [217.9 to 279.1] | 840.6 [666.2 to 1061] | 404.4 [338.6 to 483.0] | 381.1 [316.7 to 458.7]
  Final Void: number analyzed (Participants) | 105 | 41 | 44 | 56
  Final Void | 1982 [1681 to 2338] | 2051 [1561 to 2696] | 1938 [1488 to 2525] | 1729 [1368 to 2186]

11. Secondary Outcome: S-PMA (Non-Exposure Events)
Description: To measure S-phenylmercapturic acid (S-PMA, a BoExp to Benzene) in spot urine (concentration adjusted for creatinine).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS)
Number analyzed (Participants) | 77 | 32 | 32
ng/g
  Baseline: number analyzed (Participants) | 70 | 27 | 27
  Baseline | 113.2 [96.80 to 132.4] | 1441 [904.4 to 2296] | 192.6 [128.0 to 289.0]
  Final Void: number analyzed (Participants) | 71 | 22 | 31
  Final Void | 132.0 [113.7 to 153.1] | 1023 [594.5 to 1761] | 201.3 [137.5 to 294.7]

12. Secondary Outcome: S-PMA (Exposure Events)
Description: To measure S-phenylmercapturic acid (S-PMA, a BoExp to Benzene ) in spot urine (concentration adjusted for creatinine), during exposure events where some subjects used IQOS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS)
Number analyzed (Participants) | 113 | 42 | 45 | 60
ng/g
  Baseline: number analyzed (Participants) | 112 | 38 | 43 | 59
  Baseline | 123.5 [106.9 to 142.7] | 735.1 [482.9 to 1119] | 151.9 [116.9 to 197.5] | 195.3 [147.9 to 257.9]
  Final Void: number analyzed (Participants) | 111 | 41 | 44 | 58
  Final Void | 136.9 [121.4 to 154.4] | 612.5 [415.0 to 904.2] | 156.7 [124.0 to 198.1] | 229.3 [173.9 to 302.3]

13. Secondary Outcome: HEMA (Non-Exposure Events)
Description: To measure 2-hydroxyethyl mercapturic acid (HEMA, a BoExp to Ethylene Oxide) in spot urine (concentration adjusted for creatinine).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS)
Number analyzed (Participants) | 77 | 32 | 32
ng/g
  Baseline: number analyzed (Participants) | 70 | 27 | 27
  Baseline | 635.1 [540.3 to 746.5] | 1671 [1259 to 2217] | 629.1 [506.0 to 782.1]
  Final Void: number analyzed (Participants) | 70 | 22 | 29
  Final Void | 1299 [1063 to 1588] | 2595 [1819 to 3701] | 1520 [1181 to 1956]

14. Secondary Outcome: HEMA (Exposure Events)
Description: To measure 2-hydroxyethyl mercapturic acid (HEMA, a BoExp to Ethylene Oxide) in spot urine (concentration adjusted for creatinine), during exposure events where some subjects used IQOS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/g
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS)
Number analyzed (Participants) | 113 | 42 | 45 | 60
ng/g
  Baseline: number analyzed (Participants) | 112 | 38 | 43 | 59
  Baseline | 651.3 [572.1 to 741.5] | 1143 [895.6 to 1458] | 675.0 [546.2 to 834.1] | 705.0 [593.0 to 838.0]
  Final Void: number analyzed (Participants) | 105 | 41 | 44 | 56
  Final Void | 1486 [1299 to 1699] | 1967 [1547 to 2501] | 1440 [1174 to 1768] | 1513 [1270 to 1801]

15. Secondary Outcome: 3-Ethenylpyridine (3-EP) [µg/m^3]
Description: To measure IAQ, in real-time, through the assessment of concentrations of nicotine and select HPHCs representative of ETS in the air of the study site. (ISO Norm 18144:2003)
  Note that the measurements of 3-EP [µg/m^3] were below the limit of detection.
Time Frame: Measured at baseline for up to 3h prior to start of the event, then continuously during the event until 3h after the last participant has entered the event for 1h.
Measure: Number; unit: µg/m^3
Groups:
- Non-Exposure Event: For Non-Exposure Events, Indoor Air Quality measurements were performed at the Event location for up to 3h prior to the start of the Event and for 3h after the last participant has entered the Event for 1h.
- Exposure Event: For Exposure Events, Indoor Air Quality (IAQ) measurements were performed at the Event location for up to 3h prior to start of the Exposure and for 3h after the last participant had been exposed for 1h to quantify and differentiate background exposure and to assess the impact of IQOS use on IAQ.
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | NA — Below the limit of detection. | NA — Below the limit of detection.
  End of Event | NA — Below the limit of detection. | NA — Below the limit of detection.

16. Secondary Outcome: Nicotine [µg/m^3]
Description: To measure IAQ, in real-time, through the assessment of concentrations of nicotine and select HPHCs representative of ETS in the air of the study site. (ISO Norm 18144:2003)
Time Frame: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: µg/m^3
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | NA [NA to NA] — Below the limit of detection. | NA [NA to NA] — Below the limit of detection.
  End of Event | NA [NA to NA] — Below the limit of detection. | 0.9776 [0.8105 to 1.179]

17. Secondary Outcome: Acetaldehyde [µg/m^3]
Description: as for outcome 16
Time Frame: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: µg/m^3
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | 16.52 [15.50 to 17.60] | 29.20 [26.02 to 32.78]
  End of Event | 110 [91.12 to 132.8] | 187.4 [168.9 to 207.9]

18. Secondary Outcome: Acrolein [µg/m^3]
Description: as for outcome 16
Time Frame: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: µg/m^3
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | 0.03291 [0.02976 to 0.03639] | 0.07646 [0.06749 to 0.08662]
  End of Event | 0.07368 [0.05514 to 0.09845] | 0.3288 [0.2841 to 0.3805]

19. Secondary Outcome: Crotonaldehyde [µg/m^3]
Description: as for outcome 16
Time Frame: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: µg/m^3
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | 0.07621 [0.07024 to 0.08269] | 0.09775 [0.09048 to 0.1056]
  End of Event | 0.1356 [0.1167 to 0.1577] | 0.2523 [0.2335 to 0.2726]

20. Secondary Outcome: Formaldehyde [µg/m^3]
Description: as for outcome 16
Time Frame: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: µg/m^3
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | 16.60 [15.42 to 17.87] | 17.15 [16.20 to 18.16]
  End of Event | 17.49 [16.59 to 18.45] | 22.74 [21.84 to 23.67]

21. Secondary Outcome: NNN [µg/m^3]
Description: To measure IAQ, in real-time, through the assessment of concentrations of nicotine and select HPHCs representative of ETS in the air of the study site. (ISO Norm 18144:2003)
  Note that the measurements were below the limit of detection.
Time Frame: as for outcome 15
Measure: Number; unit: µg/m^3
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | NA — Below the limit of detection. | NA — Below the limit of detection.
  End of Event | NA — Below the limit of detection. | NA — Below the limit of detection.

22. Secondary Outcome: NNK [µg/m^3]
Description: To measure IAQ, in real-time, through the assessment of concentrations of nicotine and select HPHCs representative of ETS in the air of the study site. (ISO Norm 18144:2003)
  Note that the measurements of NNK [µg/m3] were below the limit of detection.
Time Frame: as for outcome 15
Measure: Number; unit: µg/m^3
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | NA — Below the limit of detection. | NA — Below the limit of detection.
  End of Event | NA — Below the limit of detection. | NA — Below the limit of detection.

23. Secondary Outcome: PM1 Particles [µg/m^3]
Description: Real-time measurements of PM1 suspended particles in air. (ISO Norm 18144:2003)
Time Frame: as for outcome 15
Measure: Mean (95% Confidence Interval); unit: µg/m^3
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | 1.489 [1.367 to 1.611] | 1.251 [1.150 to 1.353]
  End of Event | 11.508 [10.535 to 12.48] | 9.991 [9.658 to 10.325]

24. Secondary Outcome: PM2.5 Particles [µg/m^3]
Description: Real-time measurements of PM2.5 suspended particles in air. (ISO Norm 18144:2003)
Time Frame: as for outcome 15
Measure: Mean (95% Confidence Interval); unit: µg/m^3
Arm/Group | Non-Exposure Event | Exposure Event
Number analyzed (Participants) | 141 | 260
µg/m^3
  Prior to Event | 1.585 [1.460 to 1.710] | 1.340 [1.239 to 1.441]
  End of Event | 12.648 [11.568 to 13.720] | 10.755 [10.405 to 11.100]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the study, for a duration of up to 6 weeks for each subject.
Description: As this study was observational by design and was conducted in a post-market setting, adverse event (AE) reporting followed the Sponsor's already established post-market Safety Surveillance Procedures for spontaneously-reported events. In case of a medical event, the study staff were advised to call the local emergency number to ensure appropriate medical treatment. Any related cost for treatment and transportation was to be borne by the Sponsor.
Arm/Group | Non-Smokers | Cigarette Smokers | IQOS Passive Users (Not Using IQOS) | IQOS Active Users (Using IQOS)
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/74 | 0/77 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/190 | 0/74 | 0/77 | 0/60
Other Adverse Events (participants affected / at risk) | 0/190 | 0/74 | 0/77 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03550989/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT03550989/SAP_001.pdf